CLINICAL TRIAL: NCT02434289
Title: Pilot Study to Study the Feasibility and Potential Impact of a Combined Resistance Exercise and Increased Protein Intake Intervention in (Frail) Elderly People, in a Real-life Setting
Brief Title: Feasibility of a Resistance Exercise and Dietary Protein Intervention in Elderly People in Practice (ProMuscle 65PK)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Zorggroep Noordwest-Veluwe (Other); FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL51834.081.14
Record Dates: First submitted 2015-04-22; First posted 2015-05-05 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Sarcopenia
Keywords: Older adults; Dietary protein; Resistance exercise; Feasibility study; Physical functioning; Real-life setting
MeSH Terms: conditions — Sarcopenia | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistance exercise and protein products (Experimental): Practice intervention trial including resistance exercise training and intake of dietary protein products in (frail) elderly, implemented by health care professionals.
  Interventions: Dietary Supplement: Dietary protein products; Other: Resistance exercise training

INTERVENTIONS:
Dietary Supplement: Dietary protein products — Increased protein intake via dairy products, guided by a dietician.
Other: Resistance exercise training — Resistance exercise training in small groups for twelve weeks, two times a week, guided by physiotherapists.

SUMMARY:
The purpose of this pilot study is to investigate the feasibility and potential impact of a combined resistance exercise and increased protein intake intervention in (frail) elderly, in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* In home assisted (also informal care) elderly individuals, that experience loss of muscle strength
* Able to understand and perform the study procedures

Exclusion Criteria:

* Type I or type II diabetes (fasted blood glucose level ≥7,0 mmol) or hypertension, unless well regulated by medication
* Diagnosed cancer or Chronic Obstructive Pulmonary Disease (COPD)
* Severe heart failure
* Renal insufficiency (eGFR <60 mL/min/1.73 m2)
* Newly placed hip/knee prosthesis (unless fully recovered), or recent surgery (stress on scar tissue)
* Allergic or sensitive for milk proteins

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention implementation | After 12 weeks
  Feasibility includes acceptability, applicability, dose received and implementation integrity. Collected in both participants and implementing health care professionals

SECONDARY OUTCOMES:
Change in skeletal muscle mass, as measured by Dual-energy X-ray Absorptiometry (DEXA) | Baseline and 12 weeks
Change in physical performance, as measured by Short Physical performance Battery (SPPB), Timed Up-and-Go (TUG) and Six Minute Walking Test (6MWT) | Baseline and 12 weeks
Change in muscle strength, as measured by a maximum strength test | Baseline and 12 weeks
Change in Quality of life, as measured by Short-Form 36 (SF-36) | Baseline and 12 weeks
Change in Activities of Daily Living (ADL) functioning, as measured by ADL-questionnaire | Baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisette de Groot, Professor, Study Director — Wageningen University
Locations (1):
- Zorggroep Noordwest-Veluwe, locatie Randmeer, Harderwijk, Gelderland, Netherlands

REFERENCES:
- [Background] Tieland M, Dirks ML, van der Zwaluw N, Verdijk LB, van de Rest O, de Groot LC, van Loon LJ. Protein supplementation increases muscle mass gain during prolonged resistance-type exercise training in frail elderly people: a randomized, double-blind, placebo-controlled trial. J Am Med Dir Assoc. 2012 Oct;13(8):713-9. doi: 10.1016/j.jamda.2012.05.020. Epub 2012 Jul 6. PMID 22770932
- [Derived] van Dongen EJ, Leerlooijer JN, Steijns JM, Tieland M, de Groot LC, Haveman-Nies A. Translation of a tailored nutrition and resistance exercise intervention for elderly people to a real-life setting: adaptation process and pilot study. BMC Geriatr. 2017 Jan 18;17(1):25. doi: 10.1186/s12877-017-0413-8. PMID 28100190